CLINICAL TRIAL: NCT00137722
Title: Identification of Outcomes From an Asthma Disease Management Program
Brief Title: Outcomes From an Asthma Disease Management Program
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Other Study IDs: 05 08-110X
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2008-12

CONDITIONS: Asthma
Keywords: Asthma; Disease Management; Outcomes; Utilization
MeSH Terms: conditions — Asthma; Patient Acceptance of Health Care | interventions — Case Management

STUDY DESIGN:
Time Perspective: Retrospective

INTERVENTIONS:
Behavioral: Education of providers and their staff
Behavioral: Case management
Behavioral: Payment for desired behaviors

SUMMARY:
Disease management is used to manage patients who have asthma and who are enrolled in a managed care health plan. To understand the effect of disease management on asthma severity and utilization, the investigators at Children's Mercy Hospitals and Clinics, will review data from a Medicaid Health Maintenance Organization (HMO) to determine the number of health plan members with different asthma severities and what their outcomes are. This will help us to improve the service provided to these patients. The investigators wish to publish this so that other health plans can benefit from the investigators experience.

DETAILED DESCRIPTION:
Disease management is used to manage patients who have asthma and who are enrolled in a managed care health plan. To understand the effect of disease management on asthma severity and utilization, we will review data from a Medicaid HMO to determine the number of health plan members with different asthma severities and what their outcomes are. This will help us to improve the service provided to these patients.

Data on subjects already exists in the Health Management database. We will use data that has been collected between January 1, 2000 and August 18, 2005. We will use a convenience sample consisting of available subjects meeting the program criteria. The total FHP database includes approximately 50,000 members from which approximately 6,000 have been identified as having asthma.

We will create a research database that will not contain any patient-specific data. Instead, an intermediate workstation will be programmed to query the health management database and send the resulting aggregated and de-identified data to the research database for analysis on another workstation. The research database will never contain any patient identifiers nor will it contain individual patient data. It only will contain aggregated data provided by the intermediate query workstation.

Here is a complete list of variables that will be housed in the research database for subsequent analysis:

Categorical variables: Asthma severity (intermittent, mild, moderate or severe persistent), Provider office, Quarter when seen, Medication type (controller or reliever), Age category (0-4, 5-9, 10-17, >17years), active status (active or inactive), Location (ER, Inpatient, Routine visit), Case managed (yes, no), Gender, Psychosocial issues, Diagnosis (asthma, not asthma)

Continuous variables: Cost of care, Number of visits, Number of prescriptions, Number of members in the above categories, Mean Quality of life

ELIGIBILITY:
Inclusion Criteria:

* Health plan members who have undergone disease management and who have a diagnosis of asthma (ICD9 code of 493.xx)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-01; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Jay M Portnoy, MD, Principal Investigator — Children's Mercy Hospitals & Clinics
Locations (1):
- Children's Mercy Hospitals & Clinics, Kansas City, Missouri, United States